CLINICAL TRIAL: NCT01826461
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Evaluation of Twice Daily PDI-192 0.1% in Comparison to PDI-192 0.15% in the Treatment of Mild to Moderate Atopic Dermatitis in Subjects 3 Months to Less Than 18 Years of Age
Brief Title: An Evaluation of PDI-192 0.1% in Comparison to PDI-192 0.15% in the Treatment of Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PreCision Dermatology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 172-0151-202
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema; PDI-192; Precision
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PDI-192 Foam, 0.1% (Experimental): topical foam, 0.1% concentration, twice daily
  Interventions: Drug: PDI-192
- PDI-192 Foam, 0.15% (Experimental): topical foam, 0.15% concentration, twice daily
  Interventions: Drug: PDI-192
- Vehicle Foam (Placebo Comparator): topical foam, 0% concentration, twice daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: PDI-192
  Arms: PDI-192 Foam, 0.1%; PDI-192 Foam, 0.15%
Drug: Vehicle
  Arms: Vehicle Foam

SUMMARY:
This study will compare the safety and efficacy of three test article foams (PDI-192 0.1% Foam, PDI-192 0.15% Foam, and Vehicle Foam) such that a final commercial product may be selected for future development.

ELIGIBILITY:
Inclusion Criteria:

* Subject presents with a clinical diagnosis of stable mild to moderate atopic dermatitis.
* Subject has used the same type of soap, moisturizers, lotions, creams, ointments, sunscreens or other skin products, and hair products (shampoo, etc.) for at least two weeks prior to study start and agrees to continue usage with the same products and with similar frequency for the entire study.

Exclusion Criteria:

* Subject is pregnant, lactating or is planning to become pregnant during the study.
* Subject requires any topical or systemic medications or is using topical inflammatory dermatoses therapies that could affect the course of their atopic dermatitis during the study period.
* Subject has used systemic corticosteroids, immunomodulators including leukotriene inhibitors, or antimetabolites within 30 days prior to study start.
* Subject has used Ultraviolet Light Therapy (PUVA, UVB, etc.) within 30 days prior to study start.
* Subject has used topical therapies for the treatment of (or may affect) their atopic dermatitis including but not limited to corticosteroids, immunomodulators (tacrolimus, pimecrolimus, etc.), tar, calcipotriene or other vitamin D preparations, retinoids, antihistamines (doxepin, diphenhydramine, etc.), antibiotics, among others, within 14 days prior to study start.
* Subject desires excessive or prolonged exposure to ultraviolet light (e.g., sunlight, tanning beds) during the study.
* Subject has used systemic (oral, IV, etc.) antibiotic therapy within seven days prior to study start.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has used an investigational drug or investigational device treatment within 30 days prior to study start.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
"Treatment Success" based on change in Investigator's Global Assessment (IGA) | Baseline and Day 29
  Success rate, based on IGA score. Success rate is defined as the percentage of subjects who achieve "Clear" (score = 0) or "Almost Clear" (score = 1) and at least a 2-grade improvement from Baseline on the IGA score at Day 29. IGA is a measure of overall severity of atopic dermatitis using a 5-point ordinal scale from 0 = clear to 4 = severe.

SECONDARY OUTCOMES:
Change in Pruritis Severity at Day 29 | Baseline and Day 29
  Change from Baseline in the severity of pruritus (itching) at Day 29. Pruritis severity is based on a periodic subject assessment using a 4-point ordinal scale from 0 = none to 3 = severe.

OTHER OUTCOMES:
Change in Eczema Area and Severity Index (EASI) Score | Baseline and Day 29
  Percent change from Baseline in EASI scores at Day 29. EASI excludes non-key signs of eczema (such as xerosis and scaling, oozing and crusting), and subjective parameters (such as pruritus and sleep loss) in order to focus the index on key disease signs and to avoid mixing objective parameters with subjective symptoms. EASI scores range from 0 (least severe) to 72 (most severe).
Change in Body Surface Area (BSA) Affected | Baseline, Days 8, 15 and 29
  Percent change from Baseline in the percent BSA affected by disease at Days 8, 15 and 29.
Change in Clinical Signs of Atopic Dermatitis (AD) | Baseline and Days 8, 15 and 29
  Change from Baseline in severity of erythema, induration/papulation, excoriation, lichenification and oozing/crusting at Days 8, 15, and 29. All clinical signs are evaluated on a 4-point ordinal scale from 0 (none) to 3 (severe).
Change in Pruritis Severity at Days 8 and 15 | Baseline and Days 8 and 15
  Change from Baseline in the severity of pruritus (itching) at Days 8 and 15. Pruritis severity is based on a periodic subject assessment using a 4-point ordinal scale from 0 = none to 3 = severe.
Subject Assessment of Improvement in Atopic Dermatitis | Day 29
  Subject global assessment of improvement in AD at Day 29, based on a 5-point ordinal scale from 1 (excellent improvement) to 5 (worse).

CONTACTS AND LOCATIONS:
Overall Officials: Syd Dromgoole, PhD, Study Director — Therapeutics, Inc.
Locations (9):
- United States (9):
  - UCSD - Rady Children's Hospital, San Diego, California
  - Northwestern University, Chicago, Illinois
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Consulting Services, High Point, North Carolina
  - DermResearch, Inc., Austin, Texas
  - UT Houston Health Science Center, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia